CLINICAL TRIAL: NCT01118533
Title: A Prospective, Multicenter, Randomized and Single Bind Trial. Influence of Laryngoscope Blade Material on Postoperative PHARYNGEAL AND LARYNGEAL Morbidity Following Scheduled OroTracheal Intubation
Brief Title: Impact of Blades Used for Scheduled Orotracheal Intubation on Postoperative Sore Throat
Acronym: MPLIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: K080902
Record Dates: First submitted 2010-03-29; First posted 2010-05-06 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-05

CONDITIONS: Tracheal Intubation Morbidity; Sore Throat
Keywords: Intubation; Sore throat; Blades; Laryngoscopy; Morbidity
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metallic blades (Experimental): laryngoscope blade material
  Interventions: Device: metal reusable blades MacIntosh
- plastic laryngoscope blades (Active Comparator): Laryngoscope Blade Material
  Interventions: Device: Single use plastic blades HEINE XP®

INTERVENTIONS:
Device: metal reusable blades MacIntosh — laryngoscope blades
  Arms: metallic blades
Device: Single use plastic blades HEINE XP® — laryngoscope blades
  Other Names: Sign use plastic blades HEINE XP®
  Arms: plastic laryngoscope blades

SUMMARY:
Orotracheal intubation following general anesthesia requires blades to be performed. The risk of patients contamination with infectious agents related to reusable metal blades leads to promote single-use blades. Some of these latter are plastic and this material may need more strength to lift the jaw and expose the larynx before orotracheal intubation. Sometimes, change of blade, from plastic to metal, during the procedure is necessary to increase the larynx exposure. This change of blade may increase the frequency of sore throat following orotracheal intubation.

Consequently, the study hypothesis is an increase of both sore throat intensity and frequency with the plastic blades compared with the metal blades.

The primary purpose of the present study is to compare the impact of these two types of blades, metal versus plastic, on sore throat intensity and frequency following scheduled orotracheal intubation for general anesthesia

DETAILED DESCRIPTION:
Trial design :

This will be a multicenter, prospective, randomized and single-blind controlled study

Material and Methods :

The obtaining of the Ethic Committee approval allows the enrolment of 712 patients scheduled for surgery performed under general anesthesia with orotracheal intubation. Adult patients, 18 to 70 years-old, with grade I-II of ASA (American Society of Anesthesiology) status will be enrolled after clear information and obtaining, at the anesthesia visit, of the non-opposition to be enrolled in the trial.

At the anesthesia visit, the anesthesiologist will explain the purpose and protocol to the patients and then will propose them to participate to the study. The decision to be enrolled will be known at the pre-anesthesia visit, one day before the surgery. Therefore, the patients will have a delay between the anesthesia and pre-anesthesia visits to make a decision. The non-opposition to participate to the trial will be clearly mentioned in the medical file.

A randomization list will be established by a statistician. Informed and non-opposed patients will be allocated both a randomization number and a plastic or metal blade in the operating theatre via the Clean Web software.

The evaluation and measure of the primary outcome will be made in a single-blind way. The patients will evaluate the sore throat intensity being unaware of the type of blade used for the orotracheal intubation. An independent research assistant in each centre will collect data evaluated in both the operating room during the orotracheal intubation procedure and the post-operative period.

The duration of tracheal intubation will be defined as the time elapsing from the mouth insertion of the blade to the passage of the tube throughout the vocal cords announced by the operator. The intra-tracheal position of the tube will be confirmed by three squared cycles of capnography.

Protocol :

Anesthesia and monitoring:

Patients will be premedicated by hydroxyzine 1 mg kg-1 the previous evening and one hour before the transfer to the operating room.

The randomization is performed in the operating room just before the anesthesia induction.

The monitoring will be standard with:

* An electrocardiogram (lookout of cardiac rhythm modifications)
* A pulse oxymetry to lookout arterial oxygen saturation
* A non-invasive blood pressure monitoring
* A capnograph to lookout carbon dioxide elimination in the expired gas and to confirm the intra-tracheal position of the tube
* A gas analyser to control the concentration of administered halogenated volatile agents
* A neuromuscular blockade monitor to lookout the depth of the neuromuscular blockade required to perform tracheal intubation in optimal conditions. The monitoring will consist of stimulating the facial nerve 1 cm near the external eyelid corner by a train of four electric charges (30 mA). The muscular responses will be evaluated on the corrugator Supercilia by counting the number of contractions.
* A bispectral index (BIS) or entropy to monitor the hypnosis depth. The expected values will be 40-60 and 25-35, respectively.
* A manometer to control the tracheal tube cuff pressure Before anesthesia induction, patients will breathe 100% oxygen till expired oxygen concentration reach 90%. Intravenous anesthesia will be then performed with propofol (1.5-2.5 mg kg -1) as hypnotic, sufentanil (0.2 mcg kg-1) and atracurium (0.5 mg kg-1) as muscle relaxant. Cis-atracurium or vecuronium as middle acting muscle relaxant or SUNCCYNILCHOLINE as short acting muscle relaxant will be authorized. According to the randomization, the blade used for orotracheal intubation will be metal or plastic. The metal blade is reusable and the plastic blade is disposable. When the BIS or the entropy will reach 40-60 and 25-35, respectively, with efficient face mask ventilation (good thoracic amplitude following by capnography cycles), no response to the TOF at the corrugator Supercilia, the laryngoscopy will be performed according to the orotracheal intubation algorithm. Tracheal tube sizes will be 7 mm for female and 7.5 for males. Tracheal tube cuff will be standard.

After tracheal intubation, the anesthesia will be maintained with inhaled halogenated gas or intravenously. Inhaled gas will be moistened. Postoperative analgesia will be anticipated in the operating room with paracetamol 1 g, ketoprofen 100 mg and nefopam if necessary. In the absence of contraindication, the three analgesics will be administered during laparotomies. Wound and abdominal holes for laparoscopy will be infiltrated with ropivacaine. At the end of the surgery, the tracheal tube will be withdrawn according to the standard procedure recommended by the French Anesthesiology Society. Mouth secretions will be suctioned delicately. In the PACU, analgesia will be continued with according to a protocol adapted to the type of surgery. Morphine will be administered if pain VAS reaches 4/10. Pharyngeal and laryngeal morbidity evaluation will begin at the discharge of the PACU and will last 48 hours. If signs persist more than 48 hours, an ENT examination will be performed to make a diagnostic.

Statistics :

Sample size: The literature reports a 30% incidence of postoperative sore throat with metal blades. The hypothesis is that this incidence could increase from 30% to 40% if plastic blades are used. Un sample size of 356 patients per group is required to detect this increase of 10% with a Chi2 test, a statistic power (1-beta) of 0.80 and alpha type I error probability of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, 18-70 years-old scheduled for surgery planned under general anesthesia with orotracheal intubation
* Patient who has underwent a clinical examination before inclusion
* Patient who has carefully read the information notice and is not opposed to participate to the study
* Patient having a assurance policy or a similar regimen

Exclusion Criteria:

* Pregnancy
* Difficulty to understand the current language (French)
* Presence of predictive factors of difficult orotracheal intubation

  * Previous difficult tracheal intubation Grade IV of the MALLANPETI score Limited mouth opening (inter-incisive distance < 3.5 cm) Limited cervical mobility Thyromental distance < 6 cm History of radiotherapy or surgery for ENT cancer Retrognathism Presence of gastric tube for postoperative purposes Presence of Pharyngeal and Laryngeal signs before surgery
  * Type of surgery Surgery performed without orotracheal intubation Thyroid surgery ENT surgery Withdrawal of gastric banding Bariatric surgery Ambulatory surgery (one-day surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 712 (Actual)
Dates: Start 2010-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The frequency of patients presenting a post-operative sore throat whose intensity is above 4 on a visual analogue scale (VAS) graded from 0 (no pain) to 10 (unbearable pain) collected at the discharge of the post-anesthesia care unit (PACU). | Two years

SECONDARY OUTCOMES:
The frequency of patients presenting a post-operative sore throat whose intensity is different from 0/10 without swallowing | 2 years
The pain intensity will be measured at the discharge of the post-anesthesia care unit (PACU) with a slide ruler displaying a visual analogue scale graded from 0 (no pain) to 10 (unbearable pain) on the blinded face | seven days
  The pain will be evaluated everyday during two days. If the pain persists, it will be evaluated everyday till the pain disappears or till the end of the patient participation (seven days).
the degree of voice modification on a VAS | Seven days
  dysphonia
the sore throat VAS during swallowing. | seven days
  dysphagia
jaw pain | seven days
lips injuries | seven days
dental injuries | seven days
blood on the blade | seven days
the intubation difficulty score (IDS) | one day
the frequency of difficult intubation | Two years
the frequency of change of blade during the tracheal intubation procedure | two years
the tracheal intubation duration. | one day

CONTACTS AND LOCATIONS:
Overall Officials: Serge Ndoko, MD, Principal Investigator — Hospital Center of Meaux
Locations (1):
- hospital Center of Meaux, department of anesthesiology, Meaux, Meaux, France

REFERENCES:
- [Background] Amour J, Marmion F, Birenbaum A, Nicolas-Robin A, Coriat P, Riou B, Langeron O. Comparison of plastic single-use and metal reusable laryngoscope blades for orotracheal intubation during rapid sequence induction of anesthesia. Anesthesiology. 2006 Jan;104(1):60-4. doi: 10.1097/00000542-200601000-00011. PMID 16394691
- [Background] Maktabi MA, Smith RB, Todd MM. Is routine endotracheal intubation as safe as we think or wish? Anesthesiology. 2003 Aug;99(2):247-8. doi: 10.1097/00000542-200308000-00002. No abstract available. PMID 12883393